CLINICAL TRIAL: NCT03026634
Title: Prevalence and Dynamic of Sleep-disordered Breathing in Patients Pre and Post Heart Transplantation - a Prospective Single Center Trial
Brief Title: Prevalence and Dynamic of Sleep-disordered Breathing in Patients Pre and Post Heart Transplantation
Acronym: HTx-HDZ-SDB-1
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Collaborators: The German Heart Foundation (Other); Deutsche Stiftung für Herzforschung (Other)
Responsible Party: Principal Investigator, Henrik Fox, MD, Cardiologist, Heart and Diabetes Center North-Rhine Westfalia
Other Study IDs: PDSAP-HTX
Record Dates: First submitted 2016-12-14; First posted 2017-01-20 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Sleep Disordered Breathing Central; Heart Failure; Heart Transplantation
Keywords: Sleep-Disordered Breathing; Heart Failure; Heart Transplantation
MeSH Terms: conditions — Sleep Apnea, Central; Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — plasma, serum and urine samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Sleep-disordered breathing — Prevalence and dynamic of sleep-disordered breathing after heart transplantation

SUMMARY:
Sleep-disordered breathing is believed to appear at a high prevalence in end-stage heart failure patients and the presence of sleep-disordered breathing has been associated with increased mortality. This study is designed to investigate prevalence and dynamics of sleep-disordered breathing in end-stage heart failure patients pre and post heart transplantation.

DETAILED DESCRIPTION:
Sleep-disordered breathing is believed to appear at a high prevalence in end-stage heart failure patients and the presence of sleep-disordered breathing has been associated with increased mortality. This study is designed to investigate prevalence and dynamics of sleep-disordered breathing in end-stage heart failure patients pre and post heart transplantation, as this topic is hardly studied yet and previous reports suggest changes in the entity of sleep-disordered breathing through heart transplantation. The circumstances and the impact of sleep-disordered breathing or residuals in heart transplant patients is not well understood yet and will be subject of this study.

ELIGIBILITY:
Inclusion Criteria:

* End-stage heart failure patients assigned and eligible for heart transplantation

Exclusion Criteria:

* heart failure patients not eligible for heart transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage heart failure patients assigned and eligible for heart transplantation
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | 30 days after heart transplantation
  Change in Apnea Hypopnea Index (AHI /h) before and after heart transplantation

SECONDARY OUTCOMES:
Apnea Index | 30 days after heart transplantation
  Change in Apnea Index (AI /h) before and after heart transplantation
Hypopnea Index | 30 days after heart transplantation
  Change in Hypopnea Index (HI /h) before and after heart transplantation
Oxygen Desaturation Index | 30 days after heart transplantation
  Change in Oxygen Desaturation (ODI /h) before and after heart transplantation
Time SaO2 < 90 (%) | 30 days after heart transplantation
  Change in Time SaO2 < 90 (%) before and after heart transplantation
Respiration cycle length | 30 days after heart transplantation
  Change in Respiration cycle lengths before and after heart transplantation
Health Questionnaires | 30 days after heart transplantation
  Change in MLWH questionnaire, this questionnaires obtains patient's quality of life in a score (in points)
Health Questionnaires | 30 days after heart transplantation
  ESS questionnaire, this questionnaires obtains patient's sleepiness in daily life in a score (in points)
Health Questionnaires | 30 days after heart transplantation
  Short Form 12 Health Survey Questionnaire, this questionnaires obtains patient's health status in a score (in points)
Right heart catheter | 30 days after heart transplantation
  Changes in right heart catheter before and after heart transplantation
Blood gas analysis | 30 days after heart transplantation
  Changes in blood gas analyses before and after heart transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Herz- und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fox H, Puehler T, Schulz U, Bitter T, Horstkotte D, Oldenburg O. Delayed recovery from Cheyne-Stokes respiration in heart failure after successful cardiac transplantation: a case report. Transplant Proc. 2014 Sep;46(7):2462-3. doi: 10.1016/j.transproceed.2014.06.063. PMID 25242802
- [Result] Basic K, Fox H, Spiesshofer J, Bitter T, Horstkotte D, Oldenburg O. Improvements of central respiratory events, Cheyne-Stokes respiration and oxygenation in patients hospitalized for acute decompensated heart failure. Sleep Med. 2016 Nov-Dec;27-28:15-19. doi: 10.1016/j.sleep.2016.10.006. Epub 2016 Oct 28. PMID 27938912
- [Result] Oldenburg O, Wellmann B, Buchholz A, Bitter T, Fox H, Thiem U, Horstkotte D, Wegscheider K. Nocturnal hypoxaemia is associated with increased mortality in stable heart failure patients. Eur Heart J. 2016 Jun 1;37(21):1695-703. doi: 10.1093/eurheartj/ehv624. Epub 2015 Nov 26. PMID 26612581
- [Derived] Potratz M, Manukyan T, Schramm R, Costard-Jackle A, Fuchs U, Morshuis M, Guenther SPW, Rojas SV, Rudolph V, Gummert JF, Fox H. Nocturnal Hypoxemic Burden Predicts Mortality in Patients Awaiting Heart Transplantation. J Sleep Res. 2025 Nov 27:e70256. doi: 10.1111/jsr.70256. Online ahead of print. PMID 41306066